CLINICAL TRIAL: NCT01889940
Title: Effectiveness of Psycho-emotional Support in Acute Spinal Cord Injury. ESPELMA Project.
Acronym: ESPELMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ESPELMA; ESPELMA (Other Grant/Funding Number: Fundació La Marató de TV3 (ref.112910))
Record Dates: First submitted 2013-05-27; First posted 2013-07-01 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Cord Injury, Acute; Professional-Patient Relations; Sensitivity Training Groups; Patient Non-Compliance; Satisfaction
Keywords: Acute Spinal Cord Injury; Patient Satisfaction; Psychological Distress; Rehabilitation; Training Professionals; Burnout; Job Content
MeSH Terms: conditions — Spinal Cord Injuries; Patient Compliance; Personal Satisfaction; Patient Satisfaction; Burnout, Psychological | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention group. (No Intervention): The initial assessment includes pre-intervention measures (baseline) for the patient, his/her relative (or main caregiver) and the rehabilitation staff.
  Patients are assessed during the first week (or ≥ 10 days of SCI Unit admission) and at discharge (an expected average of 8 weeks). At the time of each patient's discharge, their family or main caregiver is also surveyed.
  Lastly, rehabilitation team members are also assessed across the pre-intervention phase.
- Post-intervention group. (Other): Once intervention and coaching period for professionals has ended, post-intervention sample (patients, family and professionals) is assessed with the same time criteria than the pre-intervention sample.
  Interventions: Behavioral: Training for professionals (Spinal Cord Injury Unit staff).

INTERVENTIONS:
Behavioral: Training for professionals (Spinal Cord Injury Unit staff). — Prior to the training, separate focus groups for professionals, patients & families are conducted to determine each party's needs and worries.
  Tailored training for professionals (customized according to focus groups contents) consists of 12 hours distributed in 2 days (1 day per week). It includes theoretical and practical exercises on early detection of PD, communication skills, management of psycho-emotional reactions, family interventions and teamwork alternatives. Standard motivational interviewing techniques for improving empathy skills and communication styles are employed.
  Additionally, optional on-demand small group or individual coaching sessions (after training) will be offered (50-60 minutes per session) during a 6-months period.
  Other Names: - Focus groups.; - Training.; - Coaching.
  Arms: Post-intervention group.

SUMMARY:
The purposes of the ESPELMA project are twofold: 1) To increase acute spinal cord injury patients' satisfaction with treatment while hospitalization and 2) To increase mastery among rehabilitation professionals with regard to the clinical management of patients' psychological distress.

For these purposes, a tailored training for professionals will be designed and offered.

It is hypothesized that building capacity among professionals will serve to better management of patients' distress and a greater ability to commit them to the rehabilitation process. Thus, it is expected to lead to better and faster functional recovery and consequently to higher perceived satisfaction with treatment.

DETAILED DESCRIPTION:
Background: Acute spinal cord injury leaves patients severely impaired and consequently, generates high levels of psychological distress among them and their families. This psychological distress can cause patients and their families to take a less active role in rehabilitation, which leads to lower and slower levels of functional recovery and to less perceived satisfaction with the results. In addition, rehabilitation professionals that deal with this psychological distress could ultimately experience higher stress and more risk of burnout. The aim of ESPELMA project is to train rehabilitation professionals in the clinical management of acute spinal cord injury associated psychological distress, and to measure the impact of this training on the patients' perceived satisfaction with treatment. It is hypothesized that rehabilitation professionals trained in psychological distress management will foster greater psychological well-being during hospitalization among acute spinal cord injury patients and their families, and will secure greater commitment from them to participate in the rehabilitation process. Thus, it is expected to lead to better and faster functional recovery and consequently to higher perceived satisfaction with treatment.

Methods/Design: The study follows a pre-post control group design. Participants are a sample of acute spinal cord injury patients consecutively admitted to a tertiary hospital spinal cord injury unit, their relatives, and the spinal cord injury unit staff. All participants completed a baseline survey before the intervention. Training of rehabilitation professionals comprises biweekly 6-hour sessions followed by 6-months of optional on-demand coaching. Contents of the training are customized according to focus groups. Once the training sessions end, all participants are assessed again.

Discussion: To our knowledge, no studies have yet evaluated the effectiveness of training professionals to manage psychological distress of acute spinal cord injury patients by means of motivational interviewing principles. If this training proves to be effective, several benefits could be achieved: e.g. higher job content and less burnout among professionals, as well as better patient compliance and satisfaction with treatment.

Keywords Acute Spinal Cord Injury; Patient Satisfaction; Psychological Distress; Rehabilitation; Training Professionals; Burnout; Job Content.

ELIGIBILITY:
Inclusion criteria for patients are:

* To be 15 years old or older.
* To be admitted to the SCI Unit and suffering from ASCI, regardless of neurological level cervical, thoracic, lumbar or sacral) or ASIA classification (A, B, C or D).

Exclusion criteria for patients are:

* Etiology of the injury as an acute non-traumatic SCI.
* Age younger than 15 years old and 3) Traumatic Brain Injury hampering comprehension during assessments.

One relative or main caregiver per patient is assessed.

Finally, all SCI Unit staff (rehabilitative doctors, nurses, assistant nurses, physiotherapists, physical activity instructors, the occupational therapist, social workers and hospital attendants)is also assessed.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Picker Patient Experience Questionnaire (PPE-33) | At discharge (an expected average of 8 weeks after admission).
  Satisfaction with care received, the main outcome measure of the study, is evaluated with the Spanish version of the Picker Patient Experience Questionnaire (PPE).

SECONDARY OUTCOMES:
Resilience Scale (RS-25) | At discharge (an expected average of 8 weeks after admission).
  Resilience is evaluated with the Spanish version of the Resilience Scale (RS-25).
WHOQoL-BREF (26 items) | At discharge (an expected average of 8 weeks after admission).
  Quality of life is evaluated with the WHOQOL-BREF test developed by the World Health Organization.
Biomedical and demographics | Within the first week of admission and updated at discharge (an expected average of 8 weeks after admission).
  Medical and demographical data of patients is collected according to standard procedures.
SCIM-III Questionnaire | Within the first week of admission.
  Patient functional status is measured with the third version of the Spinal Cord Independence Measure (SCIM-III) questionnaire.
ASIA Classification | Within the first week of admission.
  International Standards for Neurological Classification of SCI, developed by the American Spinal Injury Association.
HADS | Within the first week of admission (plus 7-10 days).
  Psychological distress (anxiety and depression) is evaluated using the Hospital Anxiety and Depression Scale.

OTHER OUTCOMES:
VAS for family/caregivers' satisfaction with care. | At discharge (an expected average of 8 weeks after admission); (tool for family/caregivers).
  Family/caregivers' satisfaction is assessed according to the relative who acts as the main caregiver of the patient. It is rated using a 4-point Likert scale (scoring from 1 [very unsatisfied] to 4 [very satisfied]). On open question to add any other relevant information with regard to satisfaction with care is also administered.
Resilience Scale (RS-25) | At discharge (an expected average of 8 weeks after admission); (tool for family/caregivers).
  Family/caregivers' resilience.
Jefferson Scale for Professionals Empathy (JSPE) | Baseline (during the first year of the project, months 6 to 10) and post-intervention measure (during the third year of the project, months 6 to 10); (tool for professionals).
  Rehabilitation professionals' empathy skills is rated with the Jefferson Scale for Professionals Empathy (JSPE).
Maslach Burn-out Inventory (MBI-22) | Baseline (during the first year of the project, months 6 to 10) and post-intervention measure (during the third year of the project, months 6 to 10); (tool for professionals).
  Burn-out is rated with the Maslach Burnout Inventory (MBI).
Resilience Scale (RS-25). | Baseline (during the first year of the project, months 6 to 10) and post-intervention measure (during the third year of the project, months 6 to 10); (tool for professionals).
  Resilience is evaluated with the Spanish version of the Resilience Scale (RS-25).
Job Content Questionnaire (JCQ). | Baseline (during the first year of the project, months 6 to 10) and post-intervention measure (during the third year of the project, months 6 to 10); (tool for professionals).
  Job Content was assessed with the Spanish version of the Job Content Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Lusilla-Palacios, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron de Barcelona, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Consultation-Liaison Psychiatry in a Spinal Cord Injury Unit: Theoretical Elements [Interconsulta y Psiquiatría de Enlace en una Unidad de Lesión Medular: Aspectos teóricos] Lusilla-Palacios, P., Castellano-Tejedor, C., Navarro-Marfisis, M.C., González-Viejo, M. A. Cuadernos de Medicina Psicosomática y Psiquiatría de Enlace, 2013, 106, (accepted).
- [Derived] Lusilla-Palacios P, Castellano-Tejedor C. Training a Spinal Cord Injury Rehabilitation Team in Motivational Interviewing. Rehabil Res Pract. 2015;2015:358151. doi: 10.1155/2015/358151. Epub 2015 Dec 6. PMID 26770827
- [Derived] Lusilla-Palacios P, Castellano-Tejedor C. Spinal cord injury and substance use: a systematic review. Adicciones. 2015 Dec 15;27(4):294-310. English, Spanish. PMID 26706812
- [Derived] Lusilla-Palacios P, Castellano-Tejedor C, Lucrecia-Ramirez-Garceran, Navarro-Sanchis JA, Rodriguez-Urrutia A, Parramon-Puig G, Valero-Ventura S, Cuxart-Fina A. Training professionals' communication and motivation skills to improve spinal cord injury patients' satisfaction and clinical outcomes: Study protocol of the ESPELMA trial. J Health Psychol. 2015 Oct;20(10):1357-68. doi: 10.1177/1359105313512351. Epub 2013 Dec 5. PMID 24311743